CLINICAL TRIAL: NCT00832988
Title: Comparison of in Office Interrogation vs. Remote Measurements
Brief Title: CONFIRM - Comparison of in Office Interrogation Versus Remote Measurements
Acronym: CONFIRM
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM LV001
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Pacemaker
Keywords: pacing thresholds; sensing; impedance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pacemaker patients: Patients who are implanted with a SJM Zephyr™ DR device for a standard pacing indication will be eligible
  Interventions: Other: VentricularAutoCaptureTM & ACapTM Confirm

INTERVENTIONS:
Other: VentricularAutoCaptureTM & ACapTM Confirm — The testing algorithms allow the device to display threshold measurements at time of device interrogation. These will be evaluated against manual testing results.
  Other Names: Zephyr™ pacemaker; VentricularAutoCaptureTM; ACapTM Confirm

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the automated data collection in the Zephyr device as compared to manual testing results for atrial and ventricular pacing thresholds. The secondary objectives include: to compare the in-clinic time needed to retrieve and document the automated device measurements for all tests to the additional time needed to manually measure sensing, impedance and thresholds for the same patient; to compare the accuracy of the automated device test results to manual testing results; evaluate the percentage of patients who are recommended for ACapTM Confirm utilization.

The Primary Hypotheses are:

1. The values reported from ACapTM Confirm will be within 0.125 V of the value that is obtained manually in clinic.
2. The values reported from VentricularAutoCaptureTM will be within 0.125 V of the value that is obtained manually in clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients have been implanted with their device ~ 6 months prior
* Patients must have their device evaluated at the enrolling center.
* Patients must be able to comply with the regular routine follow-up schedule of the enrolling clinic.
* Patients must be able and willing to provide written informed consent to participate in the clinical trial.
* Patients age 18 or greater.

Exclusion Criteria:

* Patient has a unipolar atrial lead implanted.
* Patients who are or may potentially be pregnant.
* Patients with persistent AF.
* Less than 1 year life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary device clinic
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of the automated data collection as compared to manual testing results for atrial and ventricular pacing thresholds | 12 and 18 months post-implant

SECONDARY OUTCOMES:
To compare the in-clinic time needed to retrieve and document the automated device measurements for all tests to the additional time needed to manually measure sensing, impedance and thresholds for the same patient. | 12 and 18 months post-implant

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Kelowna General Hospital, Kelowna, British Columbia
  - North Shore Heart Group, Vancouver, British Columbia
  - William Osler Health Centre, Brampton, Ontario
  - Peterborough Regional, Peterborough, Ontario
  - Clinique de Cardiologie Desilets, Québec, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec